CLINICAL TRIAL: NCT05412381
Title: Platelet Rich Plasma (PRP) Treatment of the Anterior Cruciate Ligament Injured Knee to Decrease the Risk of Post-traumatic Osteoarthritis (PTOA): a Randomized Double-blind Controlled Trial
Brief Title: PRP in ACLR to Prevent PTOA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0984
Record Dates: First submitted 2022-04-07; First posted 2022-06-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Injuries; Post-traumatic Osteoarthritis; PRP
Keywords: platelet-rich plasma; regenerative medicine; anterior cruciate ligament reconstruction; post-traumatic osteoarthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Injections

STUDY DESIGN:
Intervention Model Description: PRP is considered a biologic.
  We designed a double-blinded randomized controlled clinical trial with two arms:
  1. Control Arm (pre-op placebo injection, ACLR surgery + placebo injection)
  2. Investigational Arm (pre-op PRP injection, ACLR surgery + PRP injection).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Arm (Placebo Comparator): The control arm will receive a pre-op placebo injection of saline, and ACLR surgery with intra-op placebo injection
  Interventions: Procedure: placebo saline injection
- Investigational Arm (Experimental): The investigational arm will receive a pre-op PRP injection, and ACLR surgery with PRP injection
  Interventions: Procedure: platelet rich plasma (PRP) injection

INTERVENTIONS:
Procedure: platelet rich plasma (PRP) injection — We aim to evaluate early catabolic and inflammatory changes in knee joints in patients receiving PRP injections following ACL injury, as these patients are at higher risk of developing PTOA. We also aim to establish correlations between markers of biologic activity of PRP and clinical outcomes (including both patient-reported outcomes and clinical functional outcomes), with emphasis on cellular and molecular inflammatory parameters modulated by PRP.
  Other Names: Autologous Conditioned Plasma (ACP)
  Arms: Investigational Arm
Procedure: placebo saline injection — Patients randomized into the control arm will receive the placebo or saline injection
  Arms: Control Arm

SUMMARY:
The purpose of our study is to examine the effect of platelet-rich-plasma (PRP) injection on the short-term resolution of post-injury inflammation (biomarkers) and improvement in joint function in patients with acute ACL injury. This RCT has been powered based on the questionnaire KOOS Jr. but it is considered a 'pilot study' in terms of the lab analysis proposed.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury is one of the most common clinical problems among active individuals, with over 250,000 ACL reconstructions (ACLR) per year in the United States. Surgical reconstruction of the ACL is typically required in individuals who wish to return to an active lifestyle due to the presence of knee instability. The results of ACLR are predictably good as far as the ability to re-establish knee stability and to allow return to cutting and pivoting activities. However, there is a lack of effective interventions that can successfully delay or prevent the progressive degenerative changes that are known to occur following injury and that will ultimately lead to post-traumatic osteoarthritis (PTOA). PTOA accounts for nearly 12% of all cases of symptomatic OA, or approximately 5.6 million cases of lower extremity OA in the United States, carrying a cost of over $11.8 billion annually. As injury rates rise and PTOA becomes more prevalent, the associated socioeconomic burden is a significant concern since these injuries have a particularly high incidence in young adults. Many different factors likely contribute to the development of PTOA following ACLR, including the inflammatory response that occurs following injury, altered knee kinematics that can persist despite "successful" ACLR, and persistent deficits in strength of the muscles around the knee. It is well-accepted that the accumulation of inflammatory mediators and matrix degrading proteases that occurs following joint injury likely plays an important role in the initiation of the pathological process leading to PTOA. Work in animal models shows that synovial inflammation plays a central role in the development of PTOA, and studies in patients undergoing ACLR uncovered synovial fluid biomarkers with prognostic value and showed that treatment with anti-inflammatory agents modulated biomarkers of cartilage degeneration. Our preliminary RNA-seq in synovial biopsies from patients undergoing arthroscopic ACLR revealed time-dependent changes in the inflammatory gene expression profile of these tissues, further suggesting that preventative therapies that dampen inflammation early after injury and before surgery may contribute to prevent the onset of PTOA. Abnormalities in the infrapatellar fat pad (IFP) are also associated with higher inflammatory synovial fluid cytokine profile following ACL tear, highlighting the contribution of the IFP-synovial compartment to the inflammatory burden of the knee. In addition to the inflammatory response that occurs following injury, inflammation also occurs following surgery. This "double hit" may play an important role in the development of PTOA, suggesting that methods to ameliorate the inflammatory process following joint injury could represent an effective therapeutic strategy.

The current standard methods available to clinicians to treat joint inflammation include oral non-steroidal anti-inflammatory (NSAID) medications and corticosteroid injection. However, clinicians have begun to use "orthobiologics" more frequently due to their potential to diminish inflammatory and catabolic mediators while also promoting repair, and because its autologous and minimally manipulated nature is not subjected to pre-market regulatory clearance from the Food and Drug Administration. Platelet rich plasma (PRP) is a non-surgical therapy increasingly used as an alternative to NSAIDs. PRP contains and releases a wide array of bioactive molecules it has been used to treat bone, tendon, and ligament injuries, and has emerged as a potential treatment for knee osteoarthritis (OA). The currently available studies comparing intra-articular PRP injections to other means of non-surgical intervention for knee OA report promising results with the use of PRP. These data suggest that positive clinical results in OA patients are mainly related to the immune modulatory effects of PRP, dampening the intra-articular inflammatory responses.

However, the role of PRP in the treatment of knee OA remains inconclusive, largely due to inconsistencies and high variability in PRP preparations, and the limited information about the relevant components in PRP that impact clinical responses. Factors including age, sex, medical comorbidities, and genetic profile may affect the composition and biologic activity of PRP samples derived from different individuals. In addition to inter-individual variations, there is currently very little data to define how the composition and biologic activity of PRP relates to the clinical outcomes. Our recent pilot data suggests that, indeed, there are changes in composition and PRP bioactivity that may be associated with variable clinical outcomes in patients with established knee OA receiving intra-articular PRP injections. However, larger clinical trials are still required to better define these changes and to establish truly mechanistic and functional correlations. Thus, a large knowledge gap remains in our understanding of the biologically active components of PRP. Furthermore, the limited data available related to PRP and knee OA addresses treatment of established OA. There is no information available about the potential of PRP for prevention of the pathological cascade leading to PTOA.

ELIGIBILITY:
Inclusion Criteria:

* Acute ACL injury within 6 weeks of presentation
* Age 14-50
* Male or female
* Meniscus injury that can be treated with meniscectomy or repair (the lack of meniscus injury will not exclude patients)

Exclusion Criteria:

* Prior ACL reconstruction
* Prior cartilage repair procedure
* Prior meniscus surgery within 12 months
* Prior steroid, hyaluronic acid, or PRP injection within 6 months
* Other ligament injury requiring repair
* Any cartilage lesion requiring repair
* Any cartilage lesion greater than grade 2 (partial thickness injury)
* History of inflammatory arthritis or joint sepsis
* Non English speakers

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Platelet count (Thousand/uL) | Baseline
  Platelet count (Thousand/uL) will be measured by completing a complete blood count on patient's blood sample.
Platelet count (Thousand/uL) | during the procedure
  Platelet count (Thousand/uL) will be measured by completing a complete blood count on patient's blood sample.
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | Baseline
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | during the procedure
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | 2 weeks post-op
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | 6 weeks post-op
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | 6 months post-op
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | 12 months post-op
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Knee Injury and Osteoarthritis Outcome (KOOS-JR) | 24 months post-op
  This survey asks about how the patient feels about their knee. The information helps keep track of how the patient feels about their knee and how well they are able to do their usual activities.
  There is no unique measurements. Answer options per question regarding stiffness, pain, function, daily and living are: None, Mild, Moderate, Severe, and Extreme
Numeric Pain Rating Scale (NPRS) | Baseline
  This survey asks about the patient's pain levels.
  Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Numeric Pain Rating Scale (NPRS) | during the procedure
  This survey asks about the patient's pain levels.
  Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Numeric Pain Rating Scale (NPRS) | 6 weeks post-op
  This survey asks about the patient's pain levels.
  Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Numeric Pain Rating Scale (NPRS) | 6 months post-op
  This survey asks about the patient's pain levels.
  Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Numeric Pain Rating Scale (NPRS) | 12 months post-op
  This survey asks about the patient's pain levels.
  Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Numeric Pain Rating Scale (NPRS) | 24 months post-op
  This survey asks about the patient's pain levels.
  Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | Baseline
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | during the procedure
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 2 weeks post-op
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 6 weeks post-op
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 6 months post-op
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 12 months post-op
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Patient-Reported Outcomes Measurement Information System 10 (PROMIS-10) | 24 months post-op
  This survey asks about the patient's overall health and quality of life.
  Patient will be reporting on a Likert Scale formatted in the following manner for questions 1-6:
  5 = "Excellent", 4 = "Very good", 3 = "Good", 2 = "Fair", 1 = "Poor"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 7:
  5 = "Completely", 4 = "Mostly", 3 = "Moderately", 2 = "A little", 1 = "Not at all"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 8:
  1= "Never", 2 = "Rarely", 3 = "Sometimes", 4 = "Often", 5 = "Always"
  Patient will be reporting on a Likert Scale formatted in the following manner for question 9:
  1= "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe", 5 = "Very Severe"
  For question 10: Patient will be reporting a score on a scale from 0 to 10, with 0 being "No Pain" and 10 being "Worst Pain Imaginable"
Single Assessment Numeric Evaluation (SANE) | Baseline
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.
Single Assessment Numeric Evaluation (SANE) | during the procedure
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.
Single Assessment Numeric Evaluation (SANE) | 2 weeks post-op
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.
Single Assessment Numeric Evaluation (SANE) | 6 weeks post-op
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.
Single Assessment Numeric Evaluation (SANE) | 6 months post-op
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.
Single Assessment Numeric Evaluation (SANE) | 12 months post-op
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.
Single Assessment Numeric Evaluation (SANE) | 24 months post-op
  This survey asks how the patient feels about their knee.
  Patient will be reporting a percentage from 0% to 100%, with 100% being normal.

SECONDARY OUTCOMES:
Knee stability | 6 months post-surgery
  Using the KT1000 arthrometer
Knee stability | 12 months post-surgery
  Using the KT1000 arthrometer
Knee stability | 24 months post-surgery
  Using the KT1000 arthrometer
Knee strength | 6 months post-surgery
  Using the Cybex test
Knee strength | 12 months post-surgery
  Using the Cybex test
Knee strength | 24 months post-surgery
  Using the Cybex test

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/28498226/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/21884811/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/17106388/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/27145096/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/17274274/
- See also: Related information — https://daneshyari.com/article/preview/3379191.pdf?msclkid=a5e6598fc65511ecabefea898ff674d7
- See also: Related information — https://researchexperts.utmb.edu/en/publications/posttraumatic-osteoarthritis-caused-by-battlefield-injuries-the-p?msclkid=b7492b81c65511ecaa5a86702cadcdb4
- See also: Related information — https://www.semanticscholar.org/paper/Injury-Risk-Associated-With-Sports-Specialization-Field-Tepolt/13da3e2c2e558902d568c26e4a87e213c21a10e4?msclkid=caf5be44c65711ecbd93929eb70f8aa9
- See also: Related information — https://link.springer.com/content/pdf/10.1186/s12891-017-1913-6.pdf?msclkid=cb6115c6c65511ec9f779119eaa074f0
- See also: Related information — https://europepmc.org/article/PMC/PMC6076965?msclkid=d628145dc65511ec9a80c73902082d84
- See also: Related information — https://www.semanticscholar.org/paper/A-Multicenter-Study-of-Early-Anti-inflammatory-in-Lattermann-Jacobs/ef94bf8fab89b38d5e04377e2ec5c33e0d87ee53?msclkid=e3a39c2fc65511ecbb476e3f87154d88
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/31526878/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/29761471/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/28957567/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/31680217/
- See also: Related information — https://www.semanticscholar.org/paper/Proteomic-analysis-of-platelet-alpha-granules-using-Maynard-Heijnen/f494f074db92abaea4bd4cebfef75a9d67652056?msclkid=ac07be87c65711ec9e66abbbe74a81d1
- See also: Related information — https://www.semanticscholar.org/paper/Role-of-platelet-rich-plasma-in-articular-cartilage-Mascarenhas-Saltzman/1229528ee389afd977c566fc7ed3ba735e5e8ed1?msclkid=1d6518f4c65611ecaa17a90475b4fda0
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/24080861/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/20141991/
- See also: Related information — http://dryoshi.com/wp-content/uploads/2018/04/PRP-for-primary-secondary-Knee-osteoarthritis2.pdf?msclkid=365d6135c65611ecab8229d1098d131b
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/23412171/
- See also: Related information — https://www.semanticscholar.org/paper/Autologous-matrix-induced-chondrogenesis-combined-a-Dhollander-Neve/5b19a89f4fe60942a8ac7efbd40d9e13e1fa72c7?msclkid=499784f7c65611ec8665a962b68f9bb7
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/25925602/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/26831629/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/23299850/
- See also: Related information — https://pubmed.ncbi.nlm.nih.gov/27506585/
- See also: Related information — https://www.nature.com/articles/s41598-021-90174-x?msclkid=71632923c65611ecbdbbd16784373ddb